CLINICAL TRIAL: NCT01530828
Title: Immunoreactive Trypsinogen in Infants With Intestinal Perforation
Brief Title: IRT in Infants With Intestinal Perforation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Principal Investigator, Nicole Birge, Prinicpal Investigator, Children's Hospitals and Clinics of Minnesota
Other Study IDs: SPOT IRT
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Intestinal Perforation; Necrotizing Enterocolitis
Keywords: Immunoreactive Trypsinogen; Nectrotizing Enterocolitis; Premature Infants; Serial IRT
MeSH Terms: conditions — Intestinal Perforation; Enterocolitis, Necrotizing; Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Premature infants: Weight less than 1000 grams, age 1 - 16 days.

SUMMARY:
This study is designed to evaluate a novel tool to aid in the diagnosis of intestinal perforation in infants who are at high risk. Analysis of perforation rates of all infants in the three largest participating sites shows that the majority of infants with perforation will do so prior to day of life 21. This study will target the group of infants at highest risk for IP, those with birth weight less than 1000 grams, within the time frame most likely to capture the perforation. Hypothesis: An IRT value exists that can adequately differentiate premature infants with and without intestinal perforation in the first 3 weeks of life.

DETAILED DESCRIPTION:
At least 300 infants age 1-16 days will be enrolled. IRT values will be obtained daily through day of life 21, if the infant is already having labs drawn that day. The primary outcomes will be intestinal perforation and/or death on or before day of life 21. Each patient will be followed until death or discharge. Discharge will be defined as the release of the infant to home. Infants who are transferred to another NICU may be followed if the receiving NICU is one of the investigational sites. Transfer includes the release of the infant to outside units or other units within the same hospital. The purpose of this follow up is to obtain serial IRT values through day of life 21.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Birth weight less than 1000 grams
* Admitted to investigative site within first 16 days of life.

Exclusion Criteria:

* Evidence of Intestinal perforation in utero
* Suspected or confirmed custic fibrosis
* Abdominal wall defect or intestinal atresia
* Concomitant medical condition that may create an unacceptable risk.

Ages: 1 Day to 16 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Premature infants less than 1000 grams, age 1-16 days
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-09 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
To determine the onset and duration of elevation in serum IRT in infants with intestinal perforation. | 3 years

SECONDARY OUTCOMES:
Determine if factors other than intestinal perforation affect serum IRT. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospitals & Clinics of Minnesota, Saint Paul, Minnesota, United States